CLINICAL TRIAL: NCT07321249
Title: Is There an Association Between Smartsphone Addiction, Obesity and Functional Capacity in Young Adults?
Brief Title: Is There an Association Between Smartsphone Addiction and Obesity in Young Adults?
Status: Not yet recruiting | Type: Observational
Sponsor: Alaa Mohamed Naguib Ashry (Other)
Responsible Party: Sponsor-Investigator, Alaa Mohamed Naguib Ashry, lecturer of physical therapy Cairo university, Cairo University
Organization: Cairo University (Other)
Other Study IDs: No:P.TRECL/012/005821
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Obesity
Keywords: obesity; functional capacity; smartphone addiction
MeSH Terms: conditions — Obesity; Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- smartphone group

SUMMARY:
BACKGROUND: smartphone dependence causes adverse effects on one's lifestyle such as dietary habits and daily routines, resulting in overweight or obesity. Additionally, academic stress also contributes to addictive behaviors, such as smartphone addiction. Research shows that problematic smartphone use is significantly associated with loneliness, low self-esteem, and depression. Poor mental health is also proven to be a risk factor for obesity in young adults.

ELIGIBILITY:
Inclusion Criteria:

* both genders.
* Participants between the age 18 and 25 years
* Oriented, medically stable
* Sedentary lifestyle
* Use smartphone > 5 hours daily
* addiction at least 6 months before study

Exclusion Criteria:

* Patients suffering from any chronic illness (CVDS)
* Patients with neurological or musculoskeletal diseases
* Patients with kidney diseases
* Patients with liver diseases
* Diabetes
* High blood pressure
* Athletes

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: young adult
Sampling Method: Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
six minute walk test | 3 months
  a simple, self-paced test measuring how far someone can walk in six minutes on a flat surface to assess exercise capacity and cardiorespiratory function,

SECONDARY OUTCOMES:
body shape index | 3 months
  a metric for assessing a person's risk of premature death using their height, weight (mass), and waist circumference.
body shape roundness | 3 months
  Body shape roundness refers to a body type where weight is carried more in the midsection (apple shape) or describes a softer, curvier silhouette, often characterized by rounded shoulders, hips, and chest, with less definition at the waist, contrasting with more angular shapes
smartphone addiction scale | 3 months
  the scale has 10 items, each scored from 1 to 6:
  1= strongly disagree 6= strongly agree so the minimum score 10 the maximum score 60 a higher score= worse outcome, because the scale measure the smartphone addiction, and a higher score means strong symptom of addiction.
  lower score= better outcome , low score means healthier and controlled smartphone usage

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Mohamed Naguib, Lecturer, Principal Investigator — P.T. for Cardiovascular/respiratory disorders and geriatrics department Faculty of physical therapy Cairo university